CLINICAL TRIAL: NCT06964464
Title: Comparative Effectiveness of Carvedilol Versus Metoprolol Succinate in Heart Failure Patients With an Implantable Cardioverter Defibrillator
Acronym: CARVTOP-ICD
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: University of Rochester (Other)
Collaborators: Patient-Centered Outcomes Research Institute (Other)
Responsible Party: Principal Investigator, Mehmet Aktas, Associate Professor - Department of Medicine, Cardiology (SMD), University of Rochester
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: STUDY00010093; PLACER-2023C3-33489 (Other: PCORI)
Record Dates: First submitted 2025-04-30; First posted 2025-05-09 (Actual); Last update posted 2025-09-18 (Actual); Status verified 2025-09

CONDITIONS: Heart Failure With Reduced Ejection Fraction (HFrEF); Sudden Cardiac Death; Ventricular Arrhythmia; Implantable Cardioverter Defibrillator (ICD); Beta-blocker Therapy; Cardiomyopathy
Keywords: arrhythmia; heart failure; ICD; implantable cardioverter defibrillator; ICD shock; carvedilol; metoprolol succinate; beta-blocker
MeSH Terms: conditions — Death, Sudden, Cardiac; Cardiomyopathies; Arrhythmias, Cardiac; Heart Failure | interventions — Metoprolol; Carvedilol

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Metoprolol Succinate Group (Active Comparator): Participants in this group will remain on their current treatment with metoprolol succinate. The dose of metoprolol succinate may be titrated to achieve recommended target doses as per the study protocol. The aim is to assess the outcomes associated with continued use of metoprolol succinate in patients with heart failure and an implantable cardioverter defibrillator (ICD).
  Interventions: Drug: Metoprolol Succinate
- Carvedilol Group (Experimental): Participants in this group will switch from metoprolol succinate to carvedilol at an equivalent dose. The dose of carvedilol will be titrated to the recommended target dose as per the study protocol. The goal is to evaluate the comparative effectiveness of carvedilol compared to metoprolol succinate in reducing cardiovascular events in patients with heart failure and an ICD.
  Interventions: Drug: Carvedilol

INTERVENTIONS:
Drug: Metoprolol Succinate — Metoprolol succinate is a beta-blocker used for the management of heart failure with reduced ejection fraction (HFrEF). In this study, participants in the metoprolol succinate group will remain on their current treatment regimen with metoprolol succinate. The dose will be titrated to the recommended target dose as per the study protocol. The intervention aims to evaluate the effectiveness of continued use of metoprolol succinate in patients with heart failure and an implantable cardioverter defibrillator (ICD).
  Arms: Metoprolol Succinate Group
Drug: Carvedilol — Carvedilol is a non-selective beta-blocker with alpha-blocking activity used in the treatment of heart failure. In this study, participants assigned to the carvedilol group will switch from metoprolol succinate to carvedilol at an equivalent dose. The carvedilol dose will be titrated to recommended target doses according to the study protocol. This intervention aims to compare the effectiveness of carvedilol versus metoprolol succinate in improving clinical outcomes in patients with heart failure and ICDs.
  Arms: Carvedilol Group

SUMMARY:
This prospective, multicenter, open-label, randomized comparative effectiveness trial, titled CARVTOP-ICD, evaluates the impact of carvedilol versus metoprolol succinate in patients with heart failure with reduced ejection fraction (HFrEF) and an implantable cardioverter defibrillator (ICD). The study will enroll 2,000 participants across 100 U.S. sites and includes an 18-month feasibility phase with 100 participants from 15 sites. Eligible participants must be currently treated with metoprolol succinate and willing to switch to carvedilol, with randomization in a 1:1 ratio. Participants will be followed for up to 3 years, with regular assessments including ICD interrogations, medication adherence, healthcare utilization, and quality of life surveys. The primary endpoint is the first occurrence of any ICD therapy (appropriate or inappropriate), cardiovascular (CV) hospitalization, or CV death. Secondary endpoints include ICD shock burden, healthcare utilization, and patient-reported quality of life. The trial aims to provide high-quality comparative data to address clinical equipoise surrounding the two commonly used beta-blockers in HFrEF management.

DETAILED DESCRIPTION:
The Comparative Effectiveness of Carvedilol versus Metoprolol Succinate in Heart Failure Patients with an Implantable Cardioverter Defibrillator (CARVTOP-ICD) study is a prospective, multicenter, open-label, two-arm, randomized clinical trial designed to assess the comparative effectiveness of carvedilol versus metoprolol succinate in patients with heart failure with reduced ejection fraction (HFrEF) and an implantable cardioverter defibrillator (ICD). The study will enroll a total of 2,000 participants from 100 sites across the United States, with an initial feasibility phase enrolling 100 participants from 15 sites over 18 months.

The feasibility phase will assess study infrastructure, recruitment, consent processes, medication switching protocols, safety, adherence, and retention. A patient-centered approach, including engagement of caregivers and stakeholders, underpins this phase. Strategies to improve patient and provider participation, address barriers to beta-blocker switching, and ensure diversity in enrollment will be employed. Lessons learned will guide the full-scale study.

Eligible participants must have an ICD implanted for primary prevention of sudden cardiac death due to HFrEF (either ischemic or non-ischemic etiology), be currently treated with metoprolol succinate, and be willing to switch to carvedilol. Participants will be randomized 1:1 to either remain on metoprolol succinate or switch to an equivalent dose of carvedilol, with titration to maximally tolerated doses per protocol. Key exclusion criteria include treatment with any beta-blocker other than metoprolol succinate, systolic blood pressure <100 mmHg, known intolerance to carvedilol, or inability to comply with the study protocol.

The primary endpoint is the first occurrence of any ICD therapy (appropriate or inappropriate), cardiovascular hospitalization, or cardiovascular death. Secondary endpoints include the burden of ICD shocks, healthcare utilization (including emergency visits and hospitalizations), and quality of life (QoL) measured by the Kansas City Cardiomyopathy Questionnaire-12 (KCCQ-12), Florida Shock Anxiety Scale (FSAS), and Patient Health Questionnaire-2 (PHQ-2). Tertiary endpoints include specific analyses of ventricular tachyarrhythmias and atrial arrhythmias leading to inappropriate ICD therapies.

Participants will be followed for an average of 3 years. Assessments will be conducted at baseline, weeks 2 and 4, and quarterly thereafter. Study data will include standard of care tests such as cardiac imaging, ICD interrogations, laboratory measures (BNP/NT-proBNP, creatinine, BUN, potassium, sodium), NYHA classification, CV medication data, adverse events, protocol deviations, and patient-reported outcomes.

The study will also assess subgroup responses by sex, age, race/ethnicity, heart failure etiology (ischemic vs non-ischemic), ICD type (ICD vs CRT-D), and degree of LVEF impairment.

This PCORI-funded trial will generate robust, real-world evidence to guide clinical decision-making on beta-blocker choice in HFrEF patients with ICDs, addressing a significant gap in evidence and helping inform personalized treatment strategies to improve clinical and arrhythmic outcomes.

More information can be found at www.carvtop.org

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years
* ICD implanted for primary prevention for HFrEF (either ICM or NICM) with remote monitoring capability
* Current treatment with metoprolol succinate and willing to switch to carvedilol
* LVEF <50% during the past 12 months prior to consent

Exclusion Criteria:

* Unwilling or unable to follow the protocol
* Treatment with any other ßB than metoprolol succinate or no ßB treatment
* Known prior intolerance or contraindication to carvedilol
* Systolic blood pressure <100 mmHg
* Enrollment in another clinical trial
* Inability or unwilling to consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2000 (Estimated)
Dates: Start 2025-08-17 (Actual); Primary Completion 2031-06-01 (Estimated); Study Completion 2031-07-01 (Estimated)

PRIMARY OUTCOMES:
Composite Endpoint: First Occurrence of ICD Therapy, Cardiovascular Hospitalization, or Cardiovascular Death | Up to 3 years
  This composite outcome measures the time to first occurrence of one of the following events: (1) ICD therapy (appropriate or inappropriate shocks or anti-tachycardia pacing), (2) hospitalization due to cardiovascular causes, or (3) cardiovascular death. Only the first event occurring during the study period will be counted per participant.

SECONDARY OUTCOMES:
Healthcare Utilization | Average of 3 years
  Total number of the following events during the study: all-cause hospital admissions, emergency department visits, and unplanned clinic visits. All events will be captured from electronic medical records.
ICD Shock Burden | Average of 3 years
  Total number of ICD shocks (appropriate and inappropriate).
Quality of Life - Kansas City Cardiomyopathy Questionnaire-12 (KCCQ-12) | Baseline, Year 1, Year 2, Year 3
  The KCCQ-12 is a 12-item self-administered questionnaire designed to assess the health status and quality of life in patients with heart failure. It evaluates symptoms, physical and social limitations, and overall quality of life. The total score ranges from 0 to 100, with higher scores indicating better health status.
Quality of Life - Florida Shock Anxiety Scale (FSAS) | Baseline, Year 1, Year 2, Year 3
  The FSAS measures anxiety related to the possibility of receiving an ICD shock. It consists of 10 items, each rated on a 5-point Likert scale (1 = not at all, 5 = all of the time). Individual item scores are summed to produce a total score ranging from 10 to 50, with higher scores indicating greater shock-related anxiety.
Quality of Life - Patient Health Questionnaire-2 (PHQ-2) | Baseline, Year 1, Year 2, Year 3
  The PHQ-2 is a 2-item screening tool that assesses depressive symptoms, focusing on anhedonia and depressed mood over the past two weeks. Each item is scored from 0 to 3, and the total score is the sum of the two items. Higher scores indicate greater severity of depressive symptoms.

CONTACTS AND LOCATIONS:
Locations (13):
- United States (13):
  - HonorHealth, Scottsdale, Arizona
  - AdventHealth Redmond, Rome, Georgia
  - AdventHealth Shawnee Mission, Shawnee Mission, Kansas
  - Henry Ford Health System, Detroit, Michigan
  - University of Mossouri, Columbia, Missouri
  - Creighton University Medical Center, Omaha, Nebraska
  - Suny Downstate, Brooklyn, New York
  - New York-Presbyterian Brooklyn Methodist Hospital, Brooklyn, New York
  - University of Rochester Medical Center, Rochester, New York
  - CHRISTUS Trinity Mother Frances Health System, Tyler, Texas
  - Health University of Utah, Salt Lake City, Utah
  - Virginia Commonwealth University, Richmond, Virginia
  - University of Wisconsin Hospital and Clinics, Madison, Wisconsin

IPD SHARING:
Plan to Share IPD: No
Individual participant data will not be shared for this study due to privacy concerns and the need to protect patient confidentiality. We will ensure that all results are reported in aggregate form while maintaining participant anonymity.

REFERENCES:
- [Background] Packer M, Coats AJ, Fowler MB, Katus HA, Krum H, Mohacsi P, Rouleau JL, Tendera M, Castaigne A, Roecker EB, Schultz MK, DeMets DL; Carvedilol Prospective Randomized Cumulative Survival Study Group. Effect of carvedilol on survival in severe chronic heart failure. N Engl J Med. 2001 May 31;344(22):1651-8. doi: 10.1056/NEJM200105313442201. PMID 11386263
- [Background] Packer M, Bristow MR, Cohn JN, Colucci WS, Fowler MB, Gilbert EM, Shusterman NH. The effect of carvedilol on morbidity and mortality in patients with chronic heart failure. U.S. Carvedilol Heart Failure Study Group. N Engl J Med. 1996 May 23;334(21):1349-55. doi: 10.1056/NEJM199605233342101. PMID 8614419
- [Background] Poole-Wilson PA, Swedberg K, Cleland JG, Di Lenarda A, Hanrath P, Komajda M, Lubsen J, Lutiger B, Metra M, Remme WJ, Torp-Pedersen C, Scherhag A, Skene A; Carvedilol Or Metoprolol European Trial Investigators. Comparison of carvedilol and metoprolol on clinical outcomes in patients with chronic heart failure in the Carvedilol Or Metoprolol European Trial (COMET): randomised controlled trial. Lancet. 2003 Jul 5;362(9377):7-13. doi: 10.1016/S0140-6736(03)13800-7. PMID 12853193
- [Background] Diamond A, Goldenberg I, Younis A, Goldenberg I, Sampath R, Kutyifa V, Chen AY, McNitt S, Polonsky B, Steinberg JS, Zareba W, Aktas MK. Effect of Carvedilol vs Metoprolol on Atrial and Ventricular Arrhythmias Among Implantable Cardioverter-Defibrillator Recipients. JACC Clin Electrophysiol. 2023 Oct;9(10):2122-2131. doi: 10.1016/j.jacep.2023.06.009. Epub 2023 Aug 30. PMID 37656097
- [Background] Ruwald MH, Abu-Zeitone A, Jons C, Ruwald AC, McNitt S, Kutyifa V, Zareba W, Moss AJ. Impact of carvedilol and metoprolol on inappropriate implantable cardioverter-defibrillator therapy: the MADIT-CRT trial (Multicenter Automatic Defibrillator Implantation With Cardiac Resynchronization Therapy). J Am Coll Cardiol. 2013 Oct 8;62(15):1343-50. doi: 10.1016/j.jacc.2013.03.087. Epub 2013 Jun 13. PMID 23770172
- [Background] Ruwald MH, Ruwald AC, Jons C, Alexis J, McNitt S, Zareba W, Moss AJ. Effect of metoprolol versus carvedilol on outcomes in MADIT-CRT (multicenter automatic defibrillator implantation trial with cardiac resynchronization therapy). J Am Coll Cardiol. 2013 Apr 9;61(14):1518-26. doi: 10.1016/j.jacc.2013.01.020. PMID 23500269
- [Background] Fiuzat M, Wojdyla D, Kitzman D, Fleg J, Keteyian SJ, Kraus WE, Pina IL, Whellan D, O'Connor CM. Relationship of beta-blocker dose with outcomes in ambulatory heart failure patients with systolic dysfunction: results from the HF-ACTION (Heart Failure: A Controlled Trial Investigating Outcomes of Exercise Training) trial. J Am Coll Cardiol. 2012 Jul 17;60(3):208-15. doi: 10.1016/j.jacc.2012.03.023. Epub 2012 May 2. PMID 22560018